CLINICAL TRIAL: NCT03911791
Title: Screening of Helicobacter Pylori Infection in Children of Positive Infected Mothers
Brief Title: Screening of Helicobacter Pylori in Children of Positive Infected Mothers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samaa Sayed, Principle investigator, Assiut University
Other Study IDs: Prevelance of H Pylori
Record Dates: First submitted 2019-03-10; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: H Pylori Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori is aspiral shaped gram negative organism that colonized the gastric mucosa.it was showen that intra familial infection play role in transmission of H pylori and mother play the key role in transmission .

DETAILED DESCRIPTION:
Prevelance of H pylori infection in children whose mother positive infected is different according to risks factors such as mother education,work out side or not , socioeconomic status, family size and breast feeding or not.H pylori in children can be represent with recurrent abdominal pain ,recurrent diarrhea,repeated vomitting ,pallor ,fulness,non variceal hematemesis,loss of appetite,reterded growth.complication of H pylori include gastric ulcer,duodenal ulcer,gastric atrophy may lead to gastric cancer and intestinal metaplasia.

ELIGIBILITY:
Inclusion Criteria:

Child with Dyspeptic symptoms

Exclusion Criteria:

malnutrition childs Patient with metabolic disorder

Ages: 1 Day to 13 Years | Sex: All
Age Groups: Child
Study Population: Cross sectional study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess prevelance of H pylori infection in children born of infected positive mother | Period from April 2019 to April 2020
  By taken children whose mother infected ,how many of them infected by this microbe by taken these child and done the following investigastion as stool antigen test and biobsy if they are postive by test and then follow up by treatment
Asse the effect of Helicobacter pylori infection in children with anemia | Period from April 2019 to April 2020
  By knowing effect of this microbe on growth development of children by measure weigt /height through body mass index and measure heamoglbin level
  By taken children whose positive H pylori follow effect of this microbe on heamoglbin level and do investigation as complete blood count By following test such as complete blood count and heamoglbin level and if this microbe increase level of anemia or not

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Warren JR, Marshall B. Unidentified curved bacilli on gastric epithelium in active chronic gastritis. Lancet. 1983 Jun 4;1(8336):1273-5. No abstract available. PMID 6134060
- [Background] Greenberg ER, Chey WD. Defining the role of sequential therapy for H pylori infection. Lancet. 2013 Jan 19;381(9862):180-2. doi: 10.1016/S0140-6736(12)61849-2. Epub 2012 Nov 16. No abstract available. PMID 23158881